CLINICAL TRIAL: NCT06341556
Title: Zanubrutinib for Maintenance Therapy in Patients With Mantle Cell Lymphoma Who Have Remission After First-line Immunochemotherapy- a Multicenter, Prospective, Phase II Study
Brief Title: A Multicenter, Prospective, Phase II Study of Zanubrutinib for Maintenance in Patients With Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yizhen Liu, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iNHL-03
Record Dates: First submitted 2024-03-20; First posted 2024-04-02 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Mantle Cell Lymphoma; Maintenance Therapy
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): maintenance of zanubrutinib monotherapy
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Patients diagnosed with mantle cell lymphoma who have achieved remission (CR or PR) by first-line immunochemotherapy, will be treated with Zanubrutinib monotherapy for 2 years (or until PD, intolerable toxicity, death, withdrawal, or study termination).
  Other Names: Maintenance therapy with Zanubrutinib

SUMMARY:
This study aims to evaluate whether maintenance therapy with Zanubrutinib monotherapy could improve the 2-year progression free survival (PFS) of patients with mantle cell lymphoma who had remission after first-line immunochemotherapy

DETAILED DESCRIPTION:
In this study, patients diagnosed with mantle cell lymphoma who have achieved remission (CR or PR) by first-line immunochemotherapy, will be treated with Zanubrutinib monotherapy for 2 years (or until PD, intolerable toxicity, death, withdrawal, or study termination). This study aims to evaluate whether maintenance therapy with Zanubrutinib monotherapy could improve the 2-year progression free survival (PFS) of those patients, and explore the efficiency and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Histologically confirmed mantle cell lymphoma (MCL);
* Achieved complete response (CR) or partial response (PR) through first-line sufficient treatment (including immunochemotherapy with CD20 monoclonal antibody for at least 4 cycles). Frontline induction programs include but are not limited to: R-CHOP/R-DHAP, R-CHOP, BR, etc. Previous autologous hematopoietic stem cell transplantation is allowed;
* ECOG 0-2;
* Signed informed consent form;
* Having sufficient organ function: a) Hematopoietic function: Neutrophils ≥ 1.0 × 109/L, PLT ≥ 50 × 109/L, Hb ≥ 80g/L; b) Liver function: bilirubin ≤ 1.5 times the upper limit of normal (ULN), ALT and AST<3 x ULN, serum albumin ≥ 30 g/L; c) Renal function: serum Cr<1.5 × ULN, creatinine clearance rate ≥ 50mL/min (calculated according to the standard Cockcroft Gault formula, if renal dysfunction is caused by tumor compression, creatinine clearance rate ≥ 30mL/min); d) Left ventricular ejection fraction (LVEF) ≥ 50% detected by echocardiography; e) Coagulation function (unless the subject is receiving anticoagulant therapy and the coagulation parameters (PT/INR and APTT) are within the expected range of anticoagulant therapy at the time of screening): International standardized ratio (INR) ≤ 1.5 x ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 x ULN.

Exclusion Criteria:

* Individuals who are allergic to human or mouse monoclonal antibodies and have been confirmed to be allergic to Zanubrutinib capsules and/or their excipients;
* Recent major surgery (within 4 weeks prior to enrollment), excluding diagnostic surgery;
* Uncontrollable concurrent diseases (cardiovascular and cerebrovascular diseases, blood coagulation disorders, severe infectious diseases) include but are not limited to: severe acute or chronic infections requiring systemic treatment, symptomatic congestive heart failure (New York Heart Association classification III-IV) or symptomatic or poorly controlled arrhythmias Uncontrolled arterial hypertension (systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥ 100mmHg), unstable angina, active peptic ulcer, or hemorrhagic disease even after receiving standardized treatment;
* Serious accompanying diseases that interfere with conventional treatment;
* Has a history of active malignant tumors. Except for patients with skin basal cell carcinoma, superficial bladder cancer, skin squamous cell carcinoma or cervical carcinoma in situ who have received possible curative treatment and have no disease recurrence within 3 years since the start of treatment;
* Known to have active interstitial pneumonia;
* Known cases of alcohol or drug abuse;
* Active chronic hepatitis B infection (defined as HBV DNA positive): If hepatitis B virus (HBV) DNA cannot be detected during screening, patients with latent or previous hepatitis B infection (defined as positive hepatitis B surface antigen or hepatitis B core total antibody) can be included in this study. The above patients must voluntarily undergo regular HBV-DNA testing and receive appropriate antiviral treatment according to regulations. For patients with positive hepatitis C virus (HCV) antibody serological test, only when polymerase chain reaction (PCR) shows negative HCV-RNA can participate in this study.
* Patients with active HIV and syphilis infections;
* Pregnant or lactating women;
* live vaccine administered within 4 weeks prior to administering the investigational drug, inactivated virus vaccines such as for seasonal influenza are allowed;
* Continuous corticosteroid treatment currently being received, with a dose greater than 30mg/day of prednisone or equivalent medication for at least 10 days of continuous treatment;
* Suffering from active autoimmune diseases that require systematic treatment within the past 2 years (Hormone replacement therapy is not considered as a systematic treatment, such as type I diabetes, hypothyroidism patients who only need thyroid hormone replacement therapy, patients with adrenocortical or pituitary dysfunction who only need physiological dose of glucocorticoid replacement therapy can be included in the group, and patients with autoimmune diseases who do not need systematic treatment in the past 2 years can be included in the group);
* Patients with swallowing disorders who are unable to take medication orally for a long time;
* Individuals with mental disorders who affect compliance and are unable to obtain informed consent;
* The researcher determined that patients are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) | From date of patients sign informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed progression of the disease or the occurrence of death for any reason

SECONDARY OUTCOMES:
2-year event-free survival (EFS) | From date of patients sign informed consent until the date of first documented event, progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed event for any reason
overall survival | From date of patients sign informed consent until the date of death or the date of last follow-up time, whichever came first, assessed up to 2 years
  time between the date of patients sign informed consent and the date of death or the date of last follow-up time
Hematology and non hematology toxicity | Through study completion, up to 2 years.
  number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Quality of life questionnaire | Up to 2 years
  evaluate patients' quality of life by questionnaire.

OTHER OUTCOMES:
Exploratory biomarkers | Throughout the treatment period, up to 2 years
  Biomarkers for predictive factors of efficacy at baseline or during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yizhen Liu, M.D., Ph.D., Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Cancer Center, Shanghai, Shanghai Municipality